CLINICAL TRIAL: NCT00306631
Title: A Phase 2 Study of Oral MKC-1 Administered Twice Daily for 14 Consecutive Days Every 4 Weeks in Patients With Advanced or Metastatic Breast Cancer
Brief Title: A Study to Determine the Antitumor Activity and Evaluate the Safety of MKC-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Carolyn Sidor, Chief Medical Officer, Miikana Therapeutics, an EntreMed Company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-101
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: Advanced and Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MKC-1

INTERVENTIONS:
Drug: MKC-1 — Oral capsules, 30 mg and 100 mg capsule strengths; administered twice daily for 14 days in a 28 day cycle

SUMMARY:
This phase 2 study will determine the antitumor activity, based on the objective rate, of oral MKC-1, administered twice daily for 14 consecutive days every 4 weeks, in patients with advanced or metastatic breast carcinoma. The study will also evaluate the safety and response duration in patients, time to tumor progression, and overall survival in patients following MKC-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced or metastatic adenocarcinoma of the breast
* 18 years or older
* Karnofsky performance status greater than or equal to 70%
* Radiographic or physical examination evidence of at least one site of unidimensionally-measurable disease, using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Must have failed both a taxane and an anthracycline, given sequentially or in combination, either in an adjuvant or metastatic setting
* All acute toxicity of any prior chemotherapy, surgery or radiotherapy must have resolved to National Cancer Institute Common Toxicity Criteria (NCI CTC) Grade less than or equal to 1
* Lab results, within 10 days of MKC-1 administration:

  * Hemoglobin less than or equal to 9 g/dL
  * Absolute neutrophil count greater than or equal to 1.5 x 10^9/L
  * Platelet count greater than or equal to 75 x 10^9/L
  * Serum creatinine less than or equal to 1.5 x ULN (upper limit of normal)
  * AST less than or equal to 2.5 x ULN
  * Serum albumin greater than or equal to LLN (lower limit of normal)
  * Total bilirubin less than or equal to ULN
  * Alkaline phosphatase less than or equal to 2.5 x ULN
* Signed informed consent

Exclusion Criteria:

* Pre-existing hepatomegaly with disease measures greater than or equal to 2 cm below the costal margin, secondary to malignancy
* Administration of cancer specific therapy within the following periods prior to study drug initiation:

  * chemotherapy less than 3 weeks prior
  * hormonal therapy less than one week prior
  * radiation therapy less than 2 weeks prior
* Be pregnant or lactating; not employing effective birth control
* Known central nervous system (CNS) metastases unless treated, clinically stable and not requiring steroids
* Clinical evidence of bowel obstruction, active uncontrolled malabsorption syndromes or a history of total gastrectomy
* Administration of any investigational agent (therapeutic or diagnostic) within 4 weeks prior to receipt of study medication
* Uncontrolled hypercalcemia (serum calcium-corrected greater than 12 mg/dL)
* Serious cardiac condition
* Any medical conditions that, in the investigator's opinion would impose excessive risk to the patient
* Patients with previous malignancies unless free of recurrence for at least 5 years except basal cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix
* Treatment with antiretroviral therapy metabolized through CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Antitumor activity, based on the objective response rate | every 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- IUPUI, Indianapolis, Indiana, United States